CLINICAL TRIAL: NCT07313930
Title: A Single-Center, Prospective, Randomized, Controlled Study Comparing Intraoperative and Perioperative Outcomes Using the CONMED AirSeal® and Lexicon Insufflators During Laparoscopic Sleeve Gastrectomy.
Brief Title: Gastrectomy at Low Pressure Trial - (GALPT)
Acronym: GALPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SurgiQuest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DD1250901
Record Dates: First submitted 2025-12-28; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A Single-Center, Prospective, Randomized, Controlled Study Comparing Intraoperative and Perioperative Outcomes using the CONMED AirSeal® and Lexicon Insufflators during Laparoscopic Sleeve Gastrectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AirSeal® Insufflation System (AIS) (Active Comparator): Use of CONMED AirSeal® during Laparoscopic Sleeve Gastrectomy.
  Interventions: Device: AirSeal® Insufflation System (AIS)
- Lexicon Insufflator (Active Comparator): Use of Lexicon Insufflators during Laparoscopic Sleeve Gastrectomy.
  Interventions: Device: Lexicon AP 50/30 Insufflator

INTERVENTIONS:
Device: AirSeal® Insufflation System (AIS) — insufflation device used during laparoscopic sleeve gastrectomy,
  Arms: AirSeal® Insufflation System (AIS)
Device: Lexicon AP 50/30 Insufflator — insufflation device used during laparoscopic sleeve gastrectomy,
  Arms: Lexicon Insufflator

SUMMARY:
The study is designed to compare two different insufflation devices during surgery, CONMED AirSeal to Lexicon, during Laparoscopic Sleeve Gastrectomy.

DETAILED DESCRIPTION:
A Single-Center, Prospective, Randomized, Controlled Study Comparing Intraoperative and Perioperative Outcomes using the CONMED AirSeal® and Lexicon Insufflators during Laparoscopic Sleeve Gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* . Subject indicated for non-emergent sleeve gastrectomy surgery
* . Subject (or appropriate legal representatives) can provide written informed consent to participate in the study
* Male or Female aged 22 years to 65 years
* Have no significant psychopathology that could limit the subject's ability to understand the procedure, comply with medical, surgical, and/or behavioral recommendations and office visits
* Agree to refrain from any type of elective procedures that would affect body weight such as abdominal lipoplasty or liposuction, mammoplasty, or removal of excess skin for the duration of the trial.
* Are graded as American Society of Anesthesiologists (ASA) Class I, II, or III.

Exclusion Criteria:

* Subject participation in a different investigational clinical study within 90 days before screening and for the duration of this trial (unless previously approved by the investigator and Sponsor)
* Subject requiring any surgical procedure in addition to Sleeve Gastrectomy
* Previous malabsorptive or restrictive procedures performed for the treatment of obesity
* Inability to provide informed consent
* Unable or unwilling to attend follow-up visits and examinations
* Uncontrolled hypertension (≥ Systolic: 180 mmHg or Diastolic: ≥ 120 mmHg) and/or diabetes mellitus (Fasting blood sugar level: >200 mg/dL)
* Subject falls into American Society of Anesthesiologists (ASA) Class ≥ IV
* History of chronic alcohol or drug abuse within 2 years of the screening visit
* Chronic renal failure or on dialysis
* Significant complicating medical history or immunocompromise
* Subject undergoing surgery for malignant disease
* History or presence of pre-existing autoimmune connective tissue disease, e.g., systemic lupus erythematosus or scleroderma
* Immunocompromised, such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders
* Any medical condition which precludes compliance with the study
* Subject with any other clinically significant unstable medical disorder, life threatening disease, or conditions that, in the opinion of the investigator, may jeopardize the subject's well-being and/or the soundness of this clinical study or which would contra-indicate a surgical procedure
* Previous or current history of being on regular analgesia / pain killers
* Advanced refusal of blood transfusion, (if necessary)
* If female subject pregnant, planning to become pregnant within 3 months (up to 92 days of procedure), or lactating

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Pain assessment on a 0-10 numerical rating scale(NRS). | 48 hours after surgery
  Post-Operative Pain (shoulder, neck, chest and abdominal) assessment

SECONDARY OUTCOMES:
Time | 1) Evening Surgery Day- (at 8 PM) 2) Morning- (Day 1 at 8:00 AM) 3) Evening- (Day 1 at 8 PM) 4) Morning -(Day 2 at 8 AM.) 5) Evening- (Day 2 at 8 PM)
  Procedure time, recovery room time, length of stay time

CONTACTS AND LOCATIONS:
Overall Officials: Nikhilesh Sekhar, MD FACS FASMBS, Principal Investigator — Bariatric and Specialty Surgery Center of Stamford
Locations (1):
- Bariatric and Specialty Surgery Center of Stamford, Stamford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
We are looking at the aggregate statistics